CLINICAL TRIAL: NCT07260461
Title: A Multicenter, Prospective, Randomized Controlled Clinical Trial on the Efficacy and Safety of Laparoscopic Proximal Gastrectomy With Tubular Stomach-Based Right-Opening Single Flap Valvuloplasty (LPG-tbROSF) Versus Laparoscopic Total Gastrectomy for Localized Proximal Gastric Cancer.
Brief Title: The Efficacy and Safety of Laparoscopic Proximal Gastrectomy With LPG-tbROSF Versus LTG for Localized Proximal Gastric Cancer.
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: First Affiliated Hospital of Wenzhou Medical University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: KY2025-306
Record Dates: First submitted 2025-09-10; First posted 2025-12-03 (Actual); Last update posted 2025-12-03 (Actual); Status verified 2025-12

CONDITIONS: Stomach Neoplasms; Adenocarcinoma - Gastroesophageal Junction (GEJ); Gastroesophageal Junction Cancer
MeSH Terms: conditions — Stomach Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- LTG-tbROSF (Experimental): The subjects undergo laparoscopic proximal gastrectomy (LPG), with esophagogastric reconstruction performed using the right-sided overlap and single-flap valvuloplasty (ROSF) on the tubular stomach.
  Interventions: Procedure: Laparoscopic Proximal Gastrectomy with Tubular Stomach-Based Right-Opening Single Flap Valvuloplasty (LPG-tbROSF)
- LTG (Active Comparator): Patients in the control group will undergo Laparoscopic Total Gastrectomy (LTG), and digestive tract reconstruction will be performed using a standard Roux-en-Y anastomosis.
  Interventions: Procedure: Laparoscopic Proximal Gastrectomy with Tubular Stomach-Based Right-Opening Single Flap Valvuloplasty (LPG-tbROSF)

INTERVENTIONS:
Procedure: Laparoscopic Proximal Gastrectomy with Tubular Stomach-Based Right-Opening Single Flap Valvuloplasty (LPG-tbROSF) — Experimental group (tbROSF group): Participants will undergo laparoscopic proximal gastrectomy (LPG), with esophagogastric reconstruction performed using tubulized-stomach right-open single-flap valvuloplasty (tbROSF).
  Control group (LTG group): Participants will undergo laparoscopic total gastrectomy (LTG), with digestive tract reconstruction performed using a standard Roux-en-Y anastomosis.

SUMMARY:
This clinical trial is evaluating a new, function-preserving surgical technique for patients with early-stage cancer in the upper part of the stomach.

The current standard treatment is a Laparoscopic Total Gastrectomy (LTG), which involves the complete removal of the stomach. This study compares the standard LTG with an innovative procedure called Laparoscopic Proximal Gastrectomy combined with a novel anti-reflux reconstruction (LPG-tbROSF). This new technique removes only the cancerous upper portion of the stomach, aiming to preserve digestive functions and reduce post-surgery complications like acid reflux.

The main goal is to see if patients who receive the new, stomach-preserving surgery experience less body weight loss one year after the procedure compared to those who undergo the standard total gastrectomy. The research will also compare the two surgeries in terms of post-operative quality of life, nutritional status, acid reflux symptoms, safety, and long-term cancer outcomes.

The study is a multi-center, prospective, randomized controlled trial that plans to enroll 120 patients with localized cancer in the upper stomach.

ELIGIBILITY:
Inclusion Criteria:

1. Aged from 18 to 75 years old;
2. Histologically confirmed proximal gastric adenocarcinoma, CT1-2N0M0 stage;
3. The tumor was located in the proximal third of the stomach.
4. ECOG score of 0 or 1;
5. D1+ or D2 dissection according to guidelines (depending on tumor location and intraoperative evaluation).
6. ASA grade I to III;
7. The preoperative nutritional status of the patients was good without severe malnutrition.
8. Voluntarily sign informed consent.

Exclusion Criteria:

1. Concurrent with other active malignant tumors, or a history of other malignant tumors within 5 years (excluding basal cell carcinoma of the skin and carcinoma in situ of the cervix);
2. Severe cardiovascular diseases: such as NYHA class Ⅲ and above cardiac dysfunction, recent myocardial infarction (within 6 months), refractory hypertension or arrhythmia;
3. Severe respiratory diseases: severe impairment of lung function (FEV1%<50%) or chronic respiratory failure;
4. Severe liver and kidney dysfunction: ALT/AST > 3 times the upper limit of normal, or eGFR < 30 mL/min/1.73m²;
5. patients complicated with other major chronic diseases, such as active tuberculosis, rheumatoid, systemic lupus erythematosus and other autoimmune diseases that affect surgical tolerance;
6. Tumor imaging suggested the presence of distant metastasis (M1) or regional lymph node involvement, and the tumor was unresectable.
7. Complicated with other upper gastrointestinal diseases, such as active gastric ulcer, pyloric obstruction, persistent bleeding, which seriously affect the operation;
8. Previous major gastric or upper abdominal surgery (such as subtotal gastrectomy, esophagogastric anastomosis, etc.) affecting the reconstruction method;
9. Received preoperative neoadjuvant chemoradiotherapy or targeted therapy (unless specifically permitted by the study design);
10. Pregnant or lactating women;
11. Patients with mental disorders, cognitive impairment, poor compliance, inability to understand the study content, or inability to cooperate with the follow-up;
12. Severe malnutrition before surgery: BMI < 16 kg/m² or albumin < 25 g/L;
13. Other individual conditions deemed unsuitable for enrollment by the investigator (e.g., poor willingness to cooperate, high risk of loss to follow-up, etc.).

Ages: 15 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2026-01-01 (Estimated); Primary Completion 2027-09-01 (Estimated); Study Completion 2028-09-01 (Estimated)

PRIMARY OUTCOMES:
Percentage of weight loss at 12 months postoperatively | From enrollment to the end of treatment at 12 months
  Definition: The study's single primary endpoint is the percentage of body weight loss at 12 months post-operation. It is defined as the percentage decrease in a patient's body weight from the preoperative baseline to the 12-month (±7 days) postoperative follow-up.
  Objective: This endpoint serves to directly and objectively evaluate the superiority of the investigational LPG-tbROSF procedure in maintaining mid-term nutritional status compared to the standard LTG procedure.
  Formula: The calculation is performed as follows:
  Percentage of Weight Loss (%) = [ (Baseline Preoperative Weight - Postoperative 12-Month Weight) / Baseline Preoperative Weight ] × 100%.

IPD SHARING:
Plan to Share IPD: No